CLINICAL TRIAL: NCT02643238
Title: Continued Study of Artificial Vision: Evaluation of the BrainPort® System and Investigation of Visual Ambulation
Acronym: BrainPort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 111009
Record Dates: First submitted 2015-12-23; First posted 2015-12-31 (Estimated); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Blindness
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A - Blind (Experimental): Subjects will be trained to ambulate through a 40-foot obstacle course by the occupational therapy colleagues at Akron Children's Hospital after which they will be scored on their performance while using the BrainPort® system.
  Interventions: Device: BrainPort
- Group C - Control (Active Comparator): Subjects will be trained to ambulate through a 40-foot obstacle course by the occupational therapy colleagues at Akron Children's Hospital after which they will be scored on their performance while using the BrainPort® system.
  Interventions: Device: BrainPort

INTERVENTIONS:
Device: BrainPort — This system is a novel, bionic, non-invasive, vision bypass system that conveys environment images from a spectacle-frame-mounted video-camera to the brain via an electro-tactile tongue array. The electro-tactile stimulation delivered by the tongue-array placed on the tongue allows users to interpret the images of objects in their camera's visual field

SUMMARY:
The purpose of this study is to evaluate the use of an artificial vision system called Brainport system in blind patients To investigate visual, and oculomotor (eye motion) mechanisms involved in the use of the Brainport system.

DETAILED DESCRIPTION:
The prevalence of blindness in the US adult population is 0.8% and ranges from about 3/10000 to 15/10000 in children. Data from world health organization show that about 500,000 children become blind each year. The annual cost of blindness to the federal government is $4 billion and the cost of a lifetime of support and unpaid taxes for a blind person is about $1 million.

There is a need to restore vision for blind patients. Research on vision restoration develops fast. There are multiple types of approaches toward producing useful artificial vision. One of them directly sends images from a video camera to the visual cortex via an electrode array that is intracranially placed on the visual cortex of blind patients. Another one surgically places an electrode array beneath the retina for patients whose optic nerves are still healthy. Both of them require major surgery and have high risks, and neither is available for routine clinical application.

The one that is non-invasive and easy to use is called the BrainPort® system. The BrainPort® system is manufactured by Wicab, Inc. It is commercially available and affordable to any consumer. This system is a novel, bionic, non-invasive, vision bypass system that conveys environment images from a spectacle-frame-mounted video-camera to the brain via an electro-tactile tongue array. The electro-tactile stimulation delivered by the tongue-array placed on the tongue allows users to interpret the images of objects in their camera's visual field.

ELIGIBILITY:
Inclusion Criteria:

* Less than 25 years of age and be able to cooperate for full study protocol
* Have a clinical diagnosis of blindness (light perception or worse), or 20/20 vision corrected or otherwise.
* Have completed a complete ophthalmic evaluation.
* Patients recruited must be able to undergo the training to use the BrainPort® system.
* Sign informed consent (family) or assent (patient).

Exclusion Criteria:

* Have any neurologic disease, developmental delay, congenital genetic syndromes, congenital organ malformation, malformation syndromes or metabolic disease.
* Be on any medications known to affect the visual system

Ages: 10 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Average Time to completion of obstacle path (over 25 trials) in seconds | 1 month
  To evaluate the usefulness of an artificial vision system called BrainPort® system in blind patients

SECONDARY OUTCOMES:
Average Number of errors during each trial (over 25 trials) | 1 month
  To investigate the visual mechanisms underlying how the visual sensory system is involved in information processing in the presence of tongue stimulation using sensory and visually evoked potentials

CONTACTS AND LOCATIONS:
Overall Officials: Richard Hertle, MD, Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Normann RA, Maynard EM, Rousche PJ, Warren DJ. A neural interface for a cortical vision prosthesis. Vision Res. 1999 Jul;39(15):2577-87. doi: 10.1016/s0042-6989(99)00040-1. PMID 10396626
- [Background] Chowdhury V, Morley JW, Coroneo MT. Surface stimulation of the brain with a prototype array for a visual cortex prosthesis. J Clin Neurosci. 2004 Sep;11(7):750-5. doi: 10.1016/j.jocn.2003.12.010. PMID 15337140
- [Background] Chowdhury V, Morley JW, Coroneo MT. Stimulation of the retina with a multielectrode extraocular visual prosthesis. ANZ J Surg. 2005 Aug;75(8):697-704. doi: 10.1111/j.1445-2197.2005.03498.x. PMID 16076336
- [Background] World Health Organization. Preventing blindness in children: report of WHO/IAPB scientific meeting. Geneva: WHO, 2000. (WHO/PBL/00.77.)
- [Background] Sachs HG, Schanze T, Wilms M, Rentzos A, Brunner U, Gekeler F, Hesse L. Subretinal implantation and testing of polyimide film electrodes in cats. Graefes Arch Clin Exp Ophthalmol. 2005 May;243(5):464-8. doi: 10.1007/s00417-004-1049-x. Epub 2004 Dec 1. PMID 15578200
- [Background] Danilov Y, Tyler M. Brainport: an alternative input to the brain. J Integr Neurosci. 2005 Dec;4(4):537-50. doi: 10.1142/s0219635205000914. PMID 16385646
- [Background] Ptito M, Moesgaard SM, Gjedde A, Kupers R. Cross-modal plasticity revealed by electrotactile stimulation of the tongue in the congenitally blind. Brain. 2005 Mar;128(Pt 3):606-14. doi: 10.1093/brain/awh380. Epub 2005 Jan 5. PMID 15634727
- [Background] O'Shea, R. P., Roeber, U., & Bach, M. (2010). Evoked potentials: Vision. In E. B. Goldstein (Ed.), Encyclopedia of Perception (Vol. 1, pp. 399-400, xli). Los Angeles: Sage. ISBN 9781412940818